CLINICAL TRIAL: NCT05361694
Title: Two Biologically and Clinically Distinct Entities: Progressive Versus Stable Multiple Myeloma (MM) Precursor Conditions (TRANSFORMM)
Brief Title: Two Biologically and Clinically Distinct Entities: Progressive Versus Stable Multiple Myeloma (MM) Precursor Conditions
Acronym: TRANSFORMM
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: 20220067
Record Dates: First submitted 2022-04-29; First posted 2022-05-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with MGUS or SMM: Participants with either Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SMM) will be followed for disease progression to active multiple myeloma (MM) for up to 5 years.

SUMMARY:
The key aim of the study is to define the two biologically and clinically distinct entities: progressive versus stable myeloma precursor conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MGUS and SMM will be made in accordance with the clinical diagnostic criteria set forth by the 2014 International Myeloma Working Group (IMWG) Revised Criteria.2
2. The diagnoses will be confirmed by either serum/urine protein electrophoresis, immunofixation and light-chain assays; or immunohistochemistry analyses of the bone marrow biopsy, or a combination of these tests.
3. Age greater than or equal to 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
5. The patient must be competent to sign an informed consent form.

Exclusion Criteria:

1. A diagnosis of MM as defined as any patient with detectable M-protein in blood and/or urine, monoclonal plasma cells in the bone marrow, and evidence of end-organ damage based on the Calcium Elevation, Renal Failure, Anemia, and Bone Disease (CRAB) criteria and/or myeloma-defining events.

   * Patients who have received previous therapy for MM.
   * Patients with known plasma cell or related lymphoid (e.g. lymphoplasmacytic lymphoma, Amyloid Light chain (AL) amyloidosis)
2. Confirmation of pathological diagnosis is required either from the initial pathology review report or review from the UM/SCCC Hematopathologist in accordance with the clinical diagnostic criteria set forth by the International Myeloma Working Group (IMWG) or World Health Organization (WHO). Tumor tissue that has been previously collected and is available for study or that can be collected with minimal additional risk to the patient during sampling required for routine patient care or required testing on a University of Miami (UM) /Sylvester Comprehensive Cancer Center (SCCC) research protocol will be used for diagnosis.
3. Active symptomatic major organ disorder that would increase the risk of biopsy or other procedure, including but not limited to ischemic heart disease, recent myocardial infarction, active congestive heart failure, pulmonary dysfunction.

   * Active concomitant medical or psychological illnesses that may increase the risk to the patient or inability to obtain informed consent, at the discretion of the Principal Investigator.
   * Pregnant or breast-feeding women will not be eligible for any aspect of this protocol.
   * Prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with MGUS or SMM.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of progression to active Multiple Myeloma (MM) | Up to 5 years
  The rate of progression to active multiple myeloma in participants with tumors with and without myeloma defining genomic events as evaluated by treating physician via clinical assessments (including low-input DNA whole-genome sequencing)

SECONDARY OUTCOMES:
Frequency of participant conversion from MGUS/SMM to Myeloma defining genomic events | Up to 5 years
  As per treating physician evaluation of clinical assessments (including low-input DNA whole-genome sequencing)
Frequency of participant conversion from MGUS/SMM to associated progressive phenotype | Up to 5 years
  As per treating physician evaluation of clinical assessments (including low-input DNA whole-genome sequencing)
Rate of participant conversion from MGUS/SMM to Myeloma defining genomic events | Up to 5 years
  As per treating physician evaluation of clinical assessments (including low-input DNA whole-genome sequencing)
Rate of participant conversion from MGUS/SMM to associated progressive phenotype | Up to 5 years
  As per treating physician evaluation of clinical assessments (including low-input DNA whole-genome sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Landgren, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospitals, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No